CLINICAL TRIAL: NCT04619927
Title: Genotype-guided Strategy for Antithrombotic Treatment Versus Conventional Clopidogrel Therapy in Peripheral Arterial Disease.
Brief Title: Genotype-guided Strategy for Antithrombotic Treatment in Peripheral Arterial Disease.
Acronym: GENPAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Academisch Ziekenhuis Groningen (Other); Rijnstate Hospital (Other); Bernhoven Hospital (Other); Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL2020-7057
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, open label, multicenter trial.
Masking Description: This is an open label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention includes testing of patients for carriage of the CYP2C19*2 and *3 allele (loss-of-function (LOF) alleles), followed by a genotype guided antithrombotic treatment with either clopidogrel 75mg (without LOF allele, normal metabolizers), clopidogrel 150mg (one LOF allele, intermediate metabolizers), or rivaroxaban 2.5mg twice daily plus acetylsalicylic acid 100mg (two LOF alleles, poor metabolizers).
  Interventions: Genetic: Direct CYP2C19 genotyping; Drug: Poor metabolisers; Drug: Intermediate metabolisers; Drug: Normal metabolisers and unknown metaboliser state
- Comparison group (Active Comparator): The comparison group will not be prescribed clopidogrel 75mg without preceding testing for carriage of the CYP2C19*2 and *3 loss-of-function alleles. CYP2C19 genotyping will be performed at the end of the study.
  Interventions: Genetic: CYP2C19 genotyping at the end of the study; Drug: Normal metabolisers and unknown metaboliser state

INTERVENTIONS:
Genetic: Direct CYP2C19 genotyping — CYP2C19 genotype will be determined by the Spartan RX CYP2C19 point-of-care system.
  Arms: Intervention group
Genetic: CYP2C19 genotyping at the end of the study — Blood-based CYP2C19 genotyping will be performed at the end of the study
  Arms: Comparison group
Drug: Poor metabolisers — Acetylsalicylic acid 100mg once daily plus rivaroxaban 2.5mg twice daily
  Arms: Intervention group
Drug: Intermediate metabolisers — Clopidogrel 75mg twice daily
  Arms: Intervention group
Drug: Normal metabolisers and unknown metaboliser state — Clopidogrel 75mg once daily

SUMMARY:
Rationale: Peripheral arterial disease (PAD) is a common presentation of atherosclerosis. For the prevention of adverse events related to arterial thrombosis in PAD patients, clopidogrel is recommended. Clopidogrel in itself is inactive and needs to be metabolized by cytochrome P450 2C19 (CYP2C19) into the active metabolite. About 30% of PAD patients receiving clopidogrel is carrying one or two CYP2C19 loss-of-function allele(s) and do not or to a limited extent convert the prodrug into its active metabolites, and are therefore at increased risk of adverse clinical events related to arterial thrombosis. We hypothesize that genotype-guided prescription of antithrombotic treatment reduces adverse clinical events related to arterial thrombosis.

Objective: The primary aim of the GENPAD study is to evaluate the ability of genotype-guided antithrombotic treatment to reduce adverse clinical events related to arterial thrombosis in PAD patients. Secondary objectives are to evaluate the ability of genotype-guided antithrombotic treatment to reduce the separate elements of the primary composite outcome and to assess the risk of clinically relevant bleedings in patients allocated to the genotype-guided antiplatelet treatment versus standard clopidogrel prescription.

Study design: A randomized, controlled, open label, multicenter trial. Study population: Patients (n=2276) with PAD consulting a vascular surgeon for diagnosis and/or treatment, receiving clopidogrel according to the guidelines.

Intervention: Testing for carriage of the CYP2C19*2 and *3 loss-of-function alleles, followed by a genotype guided antithrombotic treatment with either clopidogrel 75mg once daily (normal metabolizers), clopidogrel 75mg twice daily (intermediate metabolizers), or low-dose rivaroxaban plus acetylsalicylic acid (poor metabolizers).

Comparator: All patients receive clopidogrel 75mg once daily without pharmacogenetic guidance.

Main study parameters/endpoints: The primary combined outcome is the occurrence of adverse clinical events related to arterial thrombosis at 24 months. The occurrence of major adverse cardiovascular events, major adverse limb events, death and clinically relevant bleedings are the secondary endpoints.

DETAILED DESCRIPTION:
Rationale: Peripheral arterial disease (PAD) is a common presentation of atherosclerosis, resulting in intermittent claudication, pain at rest or gangrene. For the prevention of adverse events related to arterial thrombosis in PAD patients, clopidogrel is recommended. Clopidogrel in itself is inactive and needs to be metabolized by cytochrome P450 2C19 (CYP2C19) into the active metabolite. About 30% of PAD patients receiving clopidogrel is carrying one or two CYP2C19 loss-of-function allele(s) and do not or to a limited extent convert the prodrug into its active metabolites, and are therefore at increased risk of adverse clinical events related to arterial thrombosis and subsequent cardiovascular death. We hypothesize that genotype-guided prescription of antithrombotic treatment reduces adverse clinical events related to arterial thrombosis.

Objective: The primary aim of the GENPAD study is to evaluate the ability of genotype-guided antithrombotic treatment to reduce adverse clinical events related to arterial thrombosis in PAD patients. Adverse clinical events of interest are major adverse cardiovascular events (myocardial infarction, stroke, transient ischemic arrack), major adverse limb events (acute/chronic limb ischemia of peripheral vascular intervention including amputation) and death. Secondary objectives are to evaluate the ability of genotype-guided antithrombotic treatment to reduce the separate elements of the primary composite outcome and to assess the risk of clinically relevant bleedings in patients allocated to the genotype-guided antiplatelet treatment versus standard clopidogrel prescription. Other objectives are to evaluate cost-effectiveness, to explore health state scores and health-related quality of life between study groups and metabolizer states and to set-up a biobank.

Study design: A randomized, controlled, open label, multicenter trial. Study population: Patients (n=2276) with PAD consulting a vascular surgeon for diagnosis and/or treatment, receiving clopidogrel according to the guidelines.

Intervention: Testing for carriage of the CYP2C19*2 and *3 loss-of-function alleles, followed by a genotype guided antithrombotic treatment with either clopidogrel 75mg once daily (normal metabolizers), clopidogrel 75mg twice daily (intermediate metabolizers), or low-dose rivaroxaban plus acetylsalicylic acid (poor metabolizers).

Comparator: All patients receive clopidogrel 75mg once daily without pharmacogenetic guidance.

Main study parameters/endpoints: The primary combined outcome is the occurrence of adverse clinical events related to arterial thrombosis at 24 months. The occurrence of major adverse cardiovascular events, major adverse limb events, death and clinically relevant bleedings are the secondary endpoints. Health state, quality of life and medical consumption will be measured with validated questionnaire. Questionnaires will be used to assess which antithrombotic treatment the participant is receiving during follow-up, medication adherence and the occurrence of extramural adverse events at 6, 12, 24 and 36 months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will visit the hospital once for informed consent procedure, blood sample withdrawal and/or buccal sample collection This visit will be combined with a routine visit to the vascular surgeon or vascular laboratory. Patients might experience some discomfort while taking blood samples and buccal sample collection for a short amount of time. The follow-up of participants will range from 6 months (minimum) to 36 months (maximum). Participants are sent questionnaires at baseline and at 6, 12, 24 and 36 months, dependent on the duration of their follow-up. Completing the questionnaires will take approximately 30 minutes. Risks regarding the study are negligible and consist of the possible adverse events related to doubling the daily dose of clopidogrel or related to rivaroxaban and acetylsalicylic acid.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Obtained written informed consent
* Indication for monotherapy clopidogrel 75mg once daily
* Ankle-brachial index < 0.9 and/or toe brachial index < 0.5
* Current or previous symptoms due to insufficient vascularization of one or two lower extremities, including intermittent claudication, pain at rest and/or gangrene (Rutherford category 1-6)
* Consulting a vascular surgeon for diagnosis, treatment and/or follow-up of PAD

Exclusion Criteria:

* known CYP2C19 genotype or metabolizer state
* treated with coumarins, Non-vitamin K Oral Anti-Coagulants, unfractionated heparin, low molecular weight heparins or double antiplatelet therapy with acetylsalicylic acid and a P2Y12 inhibitor for other indications
* contraindication for clopidogrel, acetylsalicylic acid and/or rivaroxaban
* pregnant or breastfeeding women
* unable to give informed consent (including not being able to understand the Dutch language)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2276 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of participants that experienced major adverse events | 24 months
  The number of participants that experienced a major adverse cardiovascular events, major adverse limb events or death from any cause.

SECONDARY OUTCOMES:
The number of participants that experienced major adverse cardiovascular events | 24 months
  The number of participants that experienced a myocardial infarction, stroke, transient ischemic attack or cardiovascular death.
The number of participants that experienced major adverse limb events | 24 months
  The number of participants that experienced acute limb ischemia, chronic limb ischemia or peripheral vascular intervention
The number of participants that experienced major bleeding | 24 months
  The number of participants that experienced major bleeding, including: 1) fatal bleeding, 2) symptomatic bleeding into a critical organ, 3) bleeding causing a fall in hemoglobin level of 20 g L-1 (1.24 mmol L-1) or more or leading to transfusion of two or more units of whole blood or red cells, and 4) bleeding into a surgical site requiring a second intervention.
The number of participants that experienced clinically relevant bleeding | 24 months
  The number of participants that experienced clinically relevant bleeding, including bleeding that led to: 1) hospitalization (including presentation to an acute care facility without an overnight stay), 2) a physician guided medical or surgical treatment for bleeding, or 3) a change in antithrombotic treatment.

OTHER OUTCOMES:
The cost-effectiveness of a CYP2C19 genotype-guided antithrombotic treatment strategy versus standard clopidogrel treatment | 24 months
  The costs per adverse event avoided for CYP2C19 genotype-guided antithrombotic treatment strategy compared to standard clopidogrel treatment
The difference in mean health state scores | 24 months
  Health state score measured by the EuroQol five-dimensional questionnaire five-level (EQ-5D-5L) will be determined at baseline and during follow-up. Patients score five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) on 5 levels (no problems, slight problems, moderate problems, severe problems and extreme problems), resulting in a descriptive score of 5 consecutive numbers. The validated Dutch tariff for the EQ-5D-5L will convert the descriptive score to a continuous score (range -1 to 1) in which a higher value represents a better health state than a lower value..
The difference in health-related quality of life scores | 24 months
  Health-related quality of life measured by the abbreviated World Health Organization Quality of life questionnaire (WHOQoL-Bref) will be determined at baseline and during follow-up. Patients score their quality of life with 26 questions on 4 domains (physical, psychological, social relationships and environment). Each question can be answered by 1 to 5. Scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of individual items within each domain, multiplied by 4, represents the domain score (range 4 to 20). The mean of the domain scores is the health-related quality of life score (range 4 to 20).

CONTACTS AND LOCATIONS:
Overall Officials: Michiel C Warlé, PhD, Principal Investigator — Radboud University Medical Center
Locations (11):
- Netherlands (11):
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Ziekenhuis Gelderse Vallei, Ede
  - Máxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - UMC Groningen, Groningen
  - Ommelander Ziekenhuis, Groningen
  - Maastricht University Medical Center, Maastricht
  - Radboudumc, Nijmegen
  - Canisius Wilhelmina Hospital, Nijmegen
  - Bernhoven, Uden

IPD SHARING:
Plan to Share IPD: Yes
Data will be accessible through the Data Archiving and Networked Services Electronic Archiving System (DANS EASY) repository, using Dublin Cor metadata scheme
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately after publication of the main paper for at least 15 years.
Access Criteria: A steering committee, programme committee or project leader will be charged with approving data requests.